CLINICAL TRIAL: NCT05125744
Title: Effect of Positive End Expiratory Pressure on Respiratory Muscles Activity Assessed Through Ultrasound in Intubated Patient Undergoing Assisted Ventilation
Brief Title: Effect of Positive End Expiratory Pressure on Diaphragmatic Fraction Assessed Through Ultrasound in Intubated Patient Undergoing Assisted Ventilation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera di Perugia (Other)
Responsible Party: Principal Investigator, Prof Gianmaria Cammarota, Clinical Prophessor, Azienda Ospedaliera di Perugia
Other Study IDs: 4106/19
Record Dates: First submitted 2021-10-23; First posted 2021-11-18 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Assisted Ventilation; Positive End-expiratory Pressure; Diaphragm Injury
MeSH Terms: interventions — Respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assisted Ventilation — patients will be invasively ventilated in assisted mode. In all enrolled patients ventilated in assisted mode. Diaphragmatic activity will be evaluated through ultrasound (primary end point) and electrical activity of the diaphragm (optional) at stepwise decreasing of PEEP level. Also, the activity of remaining respiratory muscles will be assessed through sonography at the same levels of PEEP (secondary end point).

SUMMARY:
The investigators aim to assess the effects of positive end-expiratory pressure (PEEP) on diaphragmatic activity evaluated through ultrasound in patients admitted to intensive care unit (ICU) for acute respiratory failure (ARF) assisted via invasive mechanical ventilation in assisted mode.

DETAILED DESCRIPTION:
All adult critically ill patients admitted to intensive care unit (ICU) and undergoing invasive mechanical ventilation (IMV) for more than 24 hours with diagnosis of acute respiratory failure (ARF) will be screened.

The exclusion criteria will be : pregnancy, neuromuscular diseases, wounds or incision at the probe placement site, contraindications to diaphragmatic and abdominal wall unltrasound, contraindications to the placement of a specific nasogastric feeding tube (Electrical activity of the diaphragm catheter).

In all enrolled patients ventilated in assisted mode, diaphragmatic activity will be evaluated through ultrasound and electrical activity of the diaphragm (primary end point) at stepwise decreasing of PEEP level. Also, the activity of remaining respiratory muscles will be assessed through sonography at the same levels of PEEP (secondary end point) Across all study phases, patients will be sedated to assure a Richmond sedation Agitation Scale (RASS) score between 0 and -1.

The following data will be recorded for each positive end-expiratory pressure explored: dosage of sedative drugs, peripheral oxygen saturation (SpO2), inspired oxygen fraction (FiO2), inpiratory and expiratory tidal volume, respiratory rate, electrical activity of the diaphragm (Eadi) (optional data), lung aeration through ultrasound or electrical impedance tomography (optional), thickness of diaphragmatic, parasternal intercostal, external oblique, internal oblique and transversus abdominis, combined with the lung ultrasound score. Thickness is measured at both end-expiration and end-inspiration for each respiratory muscles, as indirect estimation of respiratory muscles effort, and calculated according to standard formula as follows: Thickening fraction (%) = (inspiratory thickness - expiratory thickness) / expiratory thickness * 100. All ultrasonographic measurements will be performed bedside with patients in semi-recument position, only on the right side , using a portable ultrasound machine equipped with a linear (7.5 - 12.0 MHz) or convex (2.0 - 4.0 MHz) probe. The same protocol will be carried out in case of non invasive ventilation application after extubation, reducing PEEP and inspiratory support

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* invasive mechanical ventilation > 48 hours

Exclusion Criteria:

* pregnancy
* neuromuscular disease
* wounds or incision at the probe placement site.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patient admitted in intensive care unit for hypoxemic acute respiratory failure, undergoing invasive mechanical ventilation for more than 48 hours and, after this time, ventilated in Assisted Ventilation, i.e., pressure support ventilation (PSV)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic thickening fraction | 20 minutes
  The fraction of diaphragmatic thickness variations expressed in percentage during a stepwise decrease in positive end-expiratory pressure (PEEP)

SECONDARY OUTCOMES:
Lung aeration | 20 minutes
  Lung ultrasound score during a stepwise decrease in positive end-expiratory pressure (PEEP)
Peripheral oxygen saturation | 20 minutes
  Reflects the grade of peripheral oxygenation expressed in percentage during a stepwise decrease in positive end-expiratory pressure (PEEP)
Electrical activity of the diaphragm (optional) | 20 minutes
  reflects the electrical activity of the diaphragm expressed in microvolts during a stepwise decrease in positive end-expiratory pressure (PEEP)
Inspired oxygen fraction | 20 minutes
  inspired oxygen fraction during a stepwise decrease in positive end-expiratory pressure (PEEP)
Expiratory Tidal volume | 20 minutes
  Expiratory Tidal volume expressed in milliliters during a stepwise decrease in positive end-expiratory pressure (PEEP)
Respiratory rate | 20 minutes
  Respiratory rate during expressed in breaths on minute ratio during a stepwise decrease in positive end-expiratory pressure (PEEP)
Accessory respiratory muscles thickening fraction | 20 minutes
  The fractions of accessory respiratory muscles thickening fraction expressed in percentage during a stepwise decrease in positive end-expiratory pressure (PEEP)

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Perugia, Perugia, Umbria, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
single patients data on motivated request to principal investigator